CLINICAL TRIAL: NCT03659812
Title: Application of Magnetic Activated Cell Sorting (MACS) of Spermatozoa in Artificial Insemination Cycles With Donor Sperm (AID)
Brief Title: Magnetic Activated Cell Sorting in Artificial Insemination With Donor Sperm
Acronym: MACSIAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vida Recoletas Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IVISEV-006-IAD
Record Dates: First submitted 2018-04-24; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Infertility
Keywords: Magnetic activated cell sorting (MACS); Artificial insemination with donor sperm (AID); Spermatozoa; Sperm
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MACS is applied to the sperm sample (Experimental): Previous to the AID technique, the sperm sample undergoes capacitation through Percoll density gradient and MACS
  Interventions: Other: MACS technique
- MACS is not applied to the sperm sample (No Intervention): Previous to the AID technique, MACS only undergoes capacitation through Percoll density gradient, but not MACS technique

INTERVENTIONS:
Other: MACS technique — MACS is a technique that allow us to tag and detect apoptotic spermatozoa. These apoptotic spermatozoa have phosphatidylserine in their membranes, so we add magnetic beads with Annexin V, which binds specifically to phosphatidylserine. The spermatozoa are then tagged and can be retained in a magnetic field, allowing us to collect just the non-apoptotic spermatozoa.
  Arms: MACS is applied to the sperm sample

SUMMARY:
The aim of this study is to analyse the efficacy of MACS technique for the selection of spermatozoa and its effects on implantation, pregnancy and miscarriage rate. This study will be performed by two IVI clinics (IVI Sevilla and IVI Madrid) with the purpose of finding new techniques that allow us to better select spermatozoa and improve the results of assisted reproduction techniques.

ELIGIBILITY:
Inclusion Criteria:

* Women who undergo artificial insemination with donor sperm
* Signing an informed consent form to participate in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | Ultrasound examination is performed 5 weeks after artificial insemination. Pregnancy rate is calculated during the phase of data analysis.
  The number of pregnancies confirmed by ultrasound divided by the number of artificial insemination cycles. Pregnancy is confirmed by ultrasound examination.
Implantation rate | The beta hCG analysis is performed 15 days after artificial insemination. Implantation rate is calculated during the phase of data analysis.
  The number of positive results of beta human chorionic gonadotropin (hCG) test divided by the number of artificial insemination cycles. Implantation is confirmed through the analysis of beta hCG in blood.
Live birth rate | Live births are assessed at delivery (end of pregnancy period). Live birth rate is calculated during the phase of data analysis
  The number of live births divided by the number of artificial insemination cycles

SECONDARY OUTCOMES:
Sperm cell concentration | This parameter is assessed when preparing the sample for artificial insemination (one hour before artificial insemination).
  Concentration of sperm cells in sperm sample before and after applying the MACS technique
Sperm cell motility | This parameter is assessed when preparing the sample for artificial insemination (one hour before artificial insemination).
  Proportion of sperm cells with progressive motility (according to World Health Organisation 2010 criteria) before and after applying the MACS technique
Sperm cell morphology | This parameter is assessed when preparing the sample for artificial insemination (one hour before artificial insemination).
  Proportion of sperm cells with normal morphology (according to World Health Organisation 2010 criteria) before and after applying the MACS technique
Sperm cells vitality | This parameter is assessed when preparing the sample for artificial insemination (one hour before artificial insemination).
  Proportion of live sperm cells before and after applying the MACS technique
Sperm sample volume | This parameter is assessed when preparing the sample for artificial insemination (one hour before artificial insemination).
  The volume of sperm obtained after masturbation

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Sevilla, Seville, Spain